CLINICAL TRIAL: NCT02319733
Title: Plaque Stabilization and Restoration of Vascular Function by Bioresorbable Vascular Scaffold in Acute Coronary Syndrome Prone Patients
Brief Title: Plaque Stabilization and Restoration by Bioresorbable Vascular Scaffold
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient eligable subjects and new data on BVS
Sponsor: Canisius-Wilhelmina Hospital (Other)
Responsible Party: Principal Investigator, M.E.R. Gomes, dr., Canisius-Wilhelmina Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013/498
Record Dates: First submitted 2014-12-14; First posted 2014-12-18 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Vulnerable Plaque

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bioresorbable vascular scaffold (Experimental): Implantation of Bioresorbable vascular scaffold in vulnerable plaques
  Interventions: Device: Bioresorbable vascular scaffold

INTERVENTIONS:
Device: Bioresorbable vascular scaffold — Implantation of Bioresorbable vascular scaffold in vulnerable plaques

SUMMARY:
The aim of the study is to assess if implantation of a bioresorbable vascular scaffold (BVS) for intermediate coronary lesions with morphological signs of vulnerable plaque in patients prone for acute coronary syndromes (ACS) will stabilize the plaque, improve natural vasomotion and increase vascular diameter.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients between the age of 18 and 80 years
* Morise Risk score of ≥9 (intermediate or high risk) but no proven ischemia (no positive troponin or ST-elevation)
* Intermediate coronary lesion on CT scan (50-70% based on CT estimate) and a plaque with at least two of the following vulnerability criteria: Napkin ring sign, positive remodeling, low attenuation and spotty calcification
* FFR negative lesion at coronary angiogram
* Vessel diameter ≥2.5 mm on visual estimate
* GFR ≥ 45mL/min/1.73m².

Exclusion Criteria:

* High calcium score on CT scan preventing adequate evaluation of the coronary lesion.
* Lesions located in a coronary vessels previously stented.
* Lesions located at a bifurcation
* lesions involving an epicardial side branch ≥2 mm in diameter by visual assessment
* the presence of thrombus or another clinically significant stenosis in the target vessel.
* Left main (>50%) or known three vessel disease.
* Patients presenting with acute myocardial infarction, unstable arrhythmias, or patients who have a left ventricular ejection fraction <30%
* Intolerance to Aspirin, Clopidogrel, Prasugrel, Ticagrelor, Heparine or Everolimus and known true anaphylaxis to prior contrast media or known bleeding diathesis or known coagulopathy.
* Planned elective surgical procedure necessitating interruption of dual antiplatelet therapy during the first 6 months after inclusion.
* History of stent thrombosis
* Malignancies or other comorbidity with a life expectancy of less than one year or that may result in protocol noncompliance
* Pregnancy (present, suspected or planned) or positive pregnancy test (in women with childbearing potential a negative pregnancy test is mandatory)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
change in plaque cumulative score of signs of vulnerability on CT | 24 months
nominal change in percent necrotic core and thin-cap fibroatheroma at VH-IVUS | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Canisuis Wilhelmina Hospital, Nijmegen, Gelderland, Netherlands